CLINICAL TRIAL: NCT01596218
Title: Phase I Trial of Brentuximab Vedotin for Steroid Refractory Acute Graft vs. Host Disease (GvHD)
Brief Title: Brentuximab Vedotin for Steroid Refractory GvHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Seagen Inc. (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-094
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Graft vs. Host Disease
Keywords: Steroid Refractory; Acute
MeSH Terms: conditions — Graft vs Host Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Treatment Arm for all participants - Brentuximab vedotin
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Starting dose is 0.6 mg/kg weekly x 3
  Other Names: SGN-35

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational drug. Phase I studies also try to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved brentuximab vedotin for the treatment of GVHD.

Currently, corticosteroids are the standard/first line of treatment for people with GVHD. However, some patients do not achieve a good response with steroids and other experience flare-ups while tapering steroid treatment. Corticosteroid treatment has also led to a weakening of the immune system. For this reason, there have been increased attempts by researchers to find other options for the treatment of Graft vs. Host Disease.

Brentuximab vedotin is a drug that is FDA approved for the treatment of certain types of cancers, like Hodgkin's lymphoma. Recent research studies have found increased levels of protein called CD30 in people with acute GVHD. Brentuximab vedotin is designed to target CD30. Researchers have never tried to target the CD30 molecule for the treatment of GVHD, but results from other research studies show that it could help slow the growth of your disease.

In this research study, we are trying to determine the safest dose of brentuximab vedotin that can be given to patients with GVHD.

DETAILED DESCRIPTION:
This study will be broken up into two parts: induction and maintenance. The induction phase will last for 28 days and the maintenance phase will last for 12 weeks.

Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have Graft vs. Host Disease, not everyone who participates in this research study will receive the same dose of the study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

The induction phase of the trial involves finding the safest dose of brentuximab vedotin. In this phase, participants will receive 3 weekly doses on days 1, 8 and 15 of the cycle. Brentuximab vedotin is administered via intravenous infusion, which means directly into the vein, over a period of about 30 minutes.

Additionally you will undergo the following tests and procedures when you come into the clinic to receive your brentuximab vedotin: physical exam, medical history, performance status, routine and research blood tests, assessment for side effects and acute/chronic GVHD.

If you are still on this study at the end of the induction phase, meaning you have had no serious side effects and your GVHD has not progressed, ou wil continue to the next phase of this study.

Participants in the maintenance phase will receive a total of 4 doses of brentuximab vedotin every 3 weeks for a total of 12 weeks. Day 1 of the maintenance phase will be the day after the 28 day induction phase ends. You will receive a dose of brentuximab vedotin via IV infusion on Day 1 of Weeks 1,4, 7 and 10. During these visits you will undergo the same tests, procedures and assessments as the induction phase.

You will have three follow up visits after your last dose of brentuximab vedotin at 6 months, 9 months and 12 months after the end of the maintenance phase. You also have the option to talk to your physician about continuing treatment with brentuximab vedotin. However, brentuximab vedotin will only be provided by the study for the 12 week maintenance period. Afterward, brentuximab vedotin will need to be covered by your insurance or paid for out of pocket.

ELIGIBILITY:
Inclusion Criteria:

* Acute GVHD
* Corticosteroid refractory

Exclusion Criteria:

* Pregnant or breastfeeding
* Requiring mechanical ventilation
* Concurrent hepatic VOD
* Have received another study agent within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Define MTD of Brentuximab Vedotin | 2 years
  To define the maximum tolerated dose (MTD) of brentuximab vedotin when given as treatment for steroid-refractory acute GVHD

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  To test the overall response rate of brentuximab vedotin when given as treatment for steroid refractory acute GVHD
Identification of Toxicities | 2 years
  To identify the toxicities associated with brentuximab vedotin when used as therapy for steroid-refractory acute GVHD
Overall Survival | 2 years
  Overall survival at 100 days, 180 days and one year after first infusion
Description of Cumulative Incidence of Chronic GVHD | 2 years
  To describe the cumulative incidence of chronic GVHD developing in patients with acute GVHD treated with brentuximab vedotin
Assessment of Levels of Soluble CD30 | 2 years
  To assess levels of soluble CD30 and surface CD30 expression on peripheral blood T-cells in patients with acute GVHD before and after the administration of brentuximab vedotin
Assessment of Steroid Dose | 2 years
  To assess dose of steroids (mg/kg/day of prednisone equivalent) at 6 and 12 months after starting therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No